CLINICAL TRIAL: NCT03809598
Title: A Targeted Approach to Examine the Influence of Maternal Psychological Stress on Newborn Brain Outcomes
Brief Title: Roo Study on Mom and Baby Well-Being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Alice Graham, Dr. Alice Graham, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R00MH111805 (NIH)
Record Dates: First submitted 2019-01-09; First posted 2019-01-18 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Maternal Psychological Distress; Prenatal Stress; Infant Development; Functional Neuroimaging; Pregnancy Related
Keywords: Infant MRI; Brain Development; MBCT; Mindfulness
MeSH Terms: interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Intervention Model Description: The study is a randomized, control trial with an intervention arm, Mindfulness Based Cognitive Therapy (MBCT) adapted for pregnant women (Dimidjian, Goodman, et al., 2016), and treatment as usual (TAU) arm. The study will be blinded to staff (except for the study coordinator(s) and interventionists), but participant blinding is not possible due to the nature of the intervention. Participants will be randomized using a stratified block design after initial eligibility determination.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Given the use of a psychotherapeutic intervention involving participation in group sessions, participants and interventionists cannot be blinded to group assignment. The study is designed to minimize the extent to which study staff, aside from interventionists and the primary Study Coordinator(s), are aware of group assignment. The Study Coordinator(s) needs to know group assignment because they will inform participants of their group assignment and will communicate with participants regarding group attendance. The Study Coordinator(s) will be the main point of contact for participants throughout the study to reduce risk of participants revealing their group assignment to other study staff. Participants will be informed that only the Study Coordinator(s) and interventionists, if applicable, are aware of their group assignment. Therefore, in order to ensure the integrity of the research study, they should refrain from discussing their group assignment with other staff members.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Based Cognitive Therapy (Experimental): MBCT adapted for pregnancy includes 8 sequential, weekly 2-hour group sessions co-led by two master's level therapists. Sessions include: 1) introducing new mindfulness skills through in-session practice, 2) reviewing mindfulness practices and troubleshooting barriers to practice, 3) reinforcing mindfulness skills through in-session practice and debriefing, 4) learning about how thoughts influence feelings and behaviors (not all sessions), 5) providing psychoeducational information to support skills, and 6) encouraging the establishment of social support. The intervention is focused on skill development through active engagement in mindfulness practices and exercises to increase awareness of thoughts, feelings and behavior in session, and assignment and review of daily home practices.
  Interventions: Behavioral: Mindfulness Based Cognitive Therapy
- Treatment as Usual (No Intervention): All participants will receive routine prenatal care from an identified medical provider, which they have initiated on their own. They will be able to engage in any services recommended by their primary medical provider or that they voluntarily initiate. For ethical reasons, they are not prohibited from engaging in any type of therapeutic, complementary, or medication treatment (after enrollment). The TAU group will be offered a delayed treatment option, after the 6 month follow-up. This will be a 2 hour mindfulness psychoeducation session, offered between 6 and 9 months postpartum. Several core mindfulness concepts included in the full MBCT curriculum will be taught and participants will complete several brief mindfulness activities.

INTERVENTIONS:
Behavioral: Mindfulness Based Cognitive Therapy — See "Mindfulness Based Cognitive Therapy (MBCT) Arm" description
  Other Names: Mindfulness Based Cognitive Therapy for Perinatal Depression
  Arms: Mindfulness Based Cognitive Therapy

SUMMARY:
This study employs a randomized controlled trial of an established intervention, Mindfulness Based Cognitive Therapy (MBCT) adapted for pregnancy, to examine effects on various aspects of maternal psychological stress during pregnancy (magnitude and trajectories of stress) and offspring brain systems integral to healthy and maladaptive emotion regulation. This study considers other potential influences on maternal stress and psychiatric symptomatology, and infant behavior and brain development. The study population is pregnant women aged 21-45, and their infants.

DETAILED DESCRIPTION:
The study will involve an online screen of potentially eligible pregnant women. If women are eligible after the online screen, they will be invited in for an in-person assessment, including cognitive testing and a diagnostic interview, to further determine eligibility. After the assessment, they will be informed of their eligibility status and, if applicable, randomized to a Mindfulness Based Cognitive Therapy (MBCT) group involving an 8-session group-based intervention or to treatment as usual (TAU) during pregnancy followed by one mindfulness psychoeducation session postpartum. Eligible participants will then be invited in for a study visit during which they will give blood, urine, and saliva samples. Participants in the MBCT group will complete questionnaires prior to the 1st group session, after the 4th session, and after the 8th/final session. Participants in the TAU group will complete the same questionnaires at equivalent time points. All participants will come in for an in-person session at 34 weeks GA, during which they will complete questionnaires, a brief clinical interview and provide blood, urine, and saliva samples again. Participants will then come in with their infant for the infant MRI scan within one month of giving birth. Study staff will collect a hair and saliva sample from the infant at this time. Participants will have a remote visit at 6 weeks postpartum, during which time they will complete questionnaires and a clinical interview. At 6 months postpartum, participants will return for their final visit, during which they will complete questionnaires and a clinical interview. Mothers and infants will also provide a hair sample at this time. Some visits will be adapted as needed to accommodate institutional requirements with regard to restrictions due to COVID-19.

ELIGIBILITY:
Pregnant Women/ Mothers:

Inclusion and exclusion criteria for pregnant women/ mothers will be determined by a combination of the initial screen and intake assessment.

Inclusion criteria include:

1. be 21-45 years old
2. be a female who is currently pregnant (8-22 weeks GA at screening)
3. fluently speak English
4. be available and physically able to attend group scheduled meetings
5. have a single gestation, and
6. have a history of an internalizing psychiatric disorder.

Exclusion criteria include:

1. Major neurological or medical condition (e.g., diabetes, MS),
2. IQ <80
3. maternal use of psychotropic medications, insulin, or any other medications that might impact the central nervous system (at the time of enrollment)
4. current diagnosis of substance use disorder, illicit drug use or nicotine use
5. diagnosis of autism, developmental disorder involving intellectual disability or a psychotic disorder
6. current major depressive episode, eating disorder or manic episode
7. current active suicidality and/or homicidally, or interpersonal violence
8. prior history of engaging in mindfulness-based psychotherapeutic interventions (e.g., MBCT, MBSR, DBT (mindfulness module))
9. pregnancy-specific medical conditions or complications including placental abnormality or other conditions requiring bed rest
10. known congenital, genetic, or neurologic disorder of the fetus (e.g., Down syndrome, fragile X)
11. uncorrectable vision or hearing impairments (including color blindness)

Infants:

Inclusion for infants to participate in MRI scan include:

1. being between 37 and 50 weeks gestational age (GA) equivalent at time of 1st scan*
2. not meeting any of the exclusion criteria below.

   * We are using GA equivalent rather than postnatal age because infants born pre-term will not be scanned prior to term equivalent (37 weeks GA). Therefore, infants who are born preterm may be older in terms of postnatal age, but will be similar to infants born at term with regard to time since conception. The time since conception is more pertinent to our measures of brain development versus postnatal age.

Exclusion criteria for infants (specifically exclusionary for MRI scan) include:

1. congenital, genetic, or neurologic disorder (e.g., Down syndrome, fragile X)
2. major neurologic disorder at birth (e.g., bacterial meningitis, epilepsy)
3. birth < 30 weeks GA
4. medical complications following birth requiring ongoing hospitalization.
5. medical complications or health problems at or following birth, which could make an MRI scan unsafe or uncomfortable

Ages: 3 Days to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 140 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Maternal Psychological Stress | Intake - 34 Weeks GA (T5)
  Maternal psychological stress will be a composite of the Perceived Stress Scale (PSS), Beck Anxiety Inventory (BAI), and Pregnancy Distress Questionnaire (PDQ) The magnitude and trajectory of maternal psychological stress will be examined.
Maternal Depression | Intake - 34 Weeks GA (T5)
  Maternal depressive symptoms will be measured using the Center for Epidemiologic Studies Depression Scale - Revised (CESD-R). The magnitude and trajectory of maternal psychological stress will be examined.

SECONDARY OUTCOMES:
Blood assay for inflammatory marker IL6 | 34 Weeks GA (T5)
  Levels of IL6 assayed from maternal blood samples. Difference in magnitude of inflammation between groups at T5 after adjusting for inflammation prior to the intervention.
Maternal Cortisol | 34 Weeks GA (T5)
  The cortisol levels obtained from participant's hair samples to assess cumulative cortisol from pre- to post-intervention.
Neonatal Resting State fMRI scan | Infant Scan (T6)
  MRI scans with neonates will occur during natural sleep. Resting state functional connectivity will be the outcome of interest.
Neonatal Structural MRI scan | Infant Scan (T6)
  MRI scans with neonates will occur during natural sleep. Neonatal subcortical brain structure volume will be the outcome of interest.
Maternal Pregnancy Specific Psychological Stress | Intake - 34 weeks (T5)
  The Prenatal Distress Questionnaire (PDQ) is a short measure designed to assess specific worries and concerns related to pregnancy.

CONTACTS AND LOCATIONS:
Overall Officials: Alice Graham, PHD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
We propose to share individual participant data in accord with the NIMH Data Archive Data Submission Agreement.
Time Frame: In accord with the NIMH Data Archive Data Submission Agreement policies we will share data on a semi-annual basis beginning 6-months after initiating data collection and through the end of the study.
Access Criteria: Data will be available through the NIMH Data Archive by following the procedures for Data Use Certification.
URL: https://data-archive.nimh.nih.gov/

REFERENCES:
- [Background] Dimidjian S, Goodman SH, Felder JN, Gallop R, Brown AP, Beck A. Staying well during pregnancy and the postpartum: A pilot randomized trial of mindfulness-based cognitive therapy for the prevention of depressive relapse/recurrence. J Consult Clin Psychol. 2016 Feb;84(2):134-45. doi: 10.1037/ccp0000068. Epub 2015 Dec 14. PMID 26654212